CLINICAL TRIAL: NCT04352088
Title: Investigation of Phenotypes, Endotypes and Immune Response Features in Allergic Airway Diseases
Brief Title: Immune Response Features in Allergic Airway Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Brigita Sitkauskiene, Prof., Head of Department of Immunology and Allergology, Lithuanian University of Health Sciences
Other Study IDs: AKTL1
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Allergic Rhinitis; Allergic Asthma
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Allergic rhinitis patients
  Interventions: Procedure: Nasal provocation test
- Allergic rhinitis and asthma patients
  Interventions: Procedure: Nasal provocation test
- Healthy individuals
  Interventions: Procedure: Nasal provocation test

INTERVENTIONS:
Procedure: Nasal provocation test — Allergen extract under controlled conditions will be applied into nasal mucous.

SUMMARY:
This study aims to investigate immune mechanisms and phenotypes and endotypes of allergic airway diseases - allergic rhinitis and allergic asthma. Pathogenesis of these diseases are not fully investigated yet. Patients with the same disease have different dominant symptoms, course of the disease and response to treatment. Moreover, there is a hypothesis about united airway disease suggesting that allergic rhinitis and allergic asthma is different manifestation of the same disease. This led to assumption of phenotypes and endotypes. This classification which still is not unified can let to prescribe personalized treatment for every patient.

ELIGIBILITY:
Inclusion Criteria:

* Hypersensitivity to house dust mites
* Allergic rhinitis with or without mild to moderate asthma

Exclusion Criteria:

* Acute or chronic infections
* Use of systemic immunosupresants (wait 1 month)
* Use of systemic or local antihistamines (wait 1 week)
* Use of intranasal steroids (wait 1 month)
* Oncological or active autoimmune diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with allergic rhinitis with or without asthma and healthy individuals for control group.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Cytokines level in nasal lavage and peripheral blood after nasal provocation test in different groups. | 2 hours
  Cytokines (IL-13, IL-10, IL-22, etc.) level will be measured by ELISA before and after nasal provocation test with house dust mites.
  Comparison between different groups.
Cytokines level in nasal lavage and peripheral blood after nasal provocation test in different groups. | 22 hours
  Cytokines (IL-13, IL-10, IL-22, etc.) level will be measured by ELISA before and after nasal provocation test with house dust mites.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No